CLINICAL TRIAL: NCT04062019
Title: Low-dose Interleukin-2 Treatment on Idiopathic Inflammatory Myopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-PHB089-04
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Myopathy
MeSH Terms: conditions — Myositis | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interleukin-2 (Experimental): low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU/m2 once every other day, for 3 months.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU/m2 once every other day, for 3 months.
  Other Names: Recombinant Human Interleukin-2

SUMMARY:
This study aims to explore the clinical and immunological efficacy of low-dose Interleukin-2 (IL-2) on idiopathic inflammatory myopathy (IIM).

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study. Adults with active IIM will be enrolled. IIM is defined as Dermatomyositis (DM) or Polymyositis (PM), meeting the Bohan & Peter (1975) diagnostic criteria for definite or probable DM or PM. One million units of Recombinant Human Interleukin-2 (rhIL-2) was administered subcutaneously every other day for 3 months. All patients were followed up for 3 months after withdraw of IL-2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at screening visits
2. Diagnostics meet the 1975 Bohan recommendations
3. Applying of glucocorticoids (≤0.5 mg/kg/d prednisone or equivalent doses of other hormones), DMARDs (eg methotrexate, hydroxychloroquine, azathioprine, morphine, Ester, leflunomide, cyclosporine, etc.) must be stable for 4 weeks and do not increase hormone doses or other immunosuppressive agents throughout the study. If the enrolled doctor plans to stop using the current immunosuppressant or glucocorticoid, the elution period needs to be followed before enrollment. Each drug needs to meet the following elution period

   * Glucocorticoid-2 weeks
   * Immunosuppressants (including methotrexate, azathioprine, cyclosporine, tacrolimus, leflunomide, mycophenolate mofetil) - 4 weeks
   * intravenous immunogloblin (IVIg) or cyclophosphamide - 2 months
   * Rituximab - 6 months
   * Other biological agents (infliximab, adalimumab, etanercept, anakinra, etc.) -12 weeks
4. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.
5. Active Disease means active skin disease or active muscle myositis. Active skin disease as defined by a CDASI score of at least 5. The active muscle myositis defined by the baseline hand muscle strength test (MMT-8) does not exceed 142/150, wtih at least 2 additional CSMs meet the criteria specified below:

   * Patients Globle Assessment, the minimum value of 10 cm visual analog scale (VAS) is 2.0 cm
   * Physicians Globle Assessment, the minimum value on the 10 cm VAS scale is 2.0 cm
   * Health Assessment Questionnaire (HAQ) Disability Index, with a minimum value of 0.25
   * At least one muscle enzyme [including creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] High, the lowest level is 1.3 x upper limit normal
   * Global Extra-muscle Disease Activity Score, with a minimum of 1.0 cm on the 10 cm VAS scale [This measure is a comprehensive assessment by the physician based on an assessment of the physique, skin, bone, gastrointestinal, lung and heart scale activity scores Myositis Disease Activity Assessment Tool (MDAAT).

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Use rituximab or other monoclonal antibodies within 6 months.
2. Received high doses of glucocorticoid (>0.5 mg/kg/d) within 1 month.
3. Serious complications: including heart failure (≥ New York Heart Association (NYHA) class III), renal insufficiency (creatinine clearance ≤ 30 ml/min), liver dysfunction (serum ALT or AST greater than three times the upper limit of normal, or total bilirubin greater than Normal upper limit)
4. Other serious, progressive or uncontrollable hematology, gastrointestinal, endocrine, pulmonary, cardiac, neurological or brain disorders (including demyelinating diseases such as multiple sclerosis).
5. Known allergies, hyperreactivity or intolerance of IL-2 or its excipients.
6. Have a serious infection needing hospitalization (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, EB virus, tuberculosis infection), or use intravenous antibiotics to treat infection in 2 months before the enrollment.
7. Chest imaging showed abnormalities in malignant tumors or current active infections (including tuberculosis) within 3 months prior to the first use of the study drug.
8. Infection with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, it is recommended to consult a doctor who has expertise in treating HIV or hepatitis C virus infection.
9. Any known history of malignancy in the past 5 years (except for non-melanoma skin cancer, non-melanoma skin cancer or cervical tumor without recurrence within 3 months after surgical cure prior to the first study preparation).
10. Uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past 3 years, may hinder the successful completion of the study.
11. Accept or expect to receive any live virus or bacterial vaccination within 3 months prior to the first injection of the study agent, during the study period, or within 4 months after the last injection of the study agent. Bacillus Calmette - Guerin (BCG) vaccine was inoculated within 12 months after screening.
12. Pregnant, lactating women (WCBP) are reluctant to use medically approved contraceptives during treatment and 12 months after treatment.
13. Men whose partners have fertility potential but are reluctant to use appropriate medically-accepted contraceptives during treatment and 12 months after the study.
14. Adolescents with DM or PM, myositis overlaps with another connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Foxp3+Treg cells: change in percentage of total lymphocytes | week 12
  Treg refers to regulatory T cells

SECONDARY OUTCOMES:
MMT-8 | week12 and 24
  MMT-8; a set of 8 designated muscles tested bilaterally [potential score 0 - 150]
CDASI activity score | week12 and 24
  The CDASI is a clinician-scored single page instrument that separately measures activity and damage in the skin of DM patients for use in clinical practice or clinical/therapeutic studies. Disease involvement in 15 different anatomical locations is rated using three activity (erythema, scale, erosion/ulceration) and two damage (poikiloderma, calcinosis) measures. The presence and severity of Gottron's papules, periungual changes and alopecia are also captured. Disease activity is scored from 0 to 100; higher scores indicate greater disease severity.
Physician's Global Disease Activity VAS | week 12 and 24
  Physician's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis).
Safety and tolerability of interleukin-2 as assessed by incidence of adverse events reported and observed | up tp 24 weeks
  we will report frequency of adverse events
Patient's Global Disease Activity VAS | week 12 and 24
  Patient's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis).
Proportion of subjects meeting the definition of improvement (DOI) | week12 and 24
  The primary outcome will be to compare the proportion of subjects meeting the definition of improvement (DOI) at visits 3 after the 3-month treatment period. The DOI for this trial is a composite utilizing the six core set measures (CSM): 3 of 6 CSM improved by ≥ 20%, with no more than 2 CSM worsening by ≥25% (a worsening measure cannot be the MMT).

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohan A, Peter JB, Bowman RL, Pearson CM. Computer-assisted analysis of 153 patients with polymyositis and dermatomyositis. Medicine (Baltimore). 1977 Jul;56(4):255-86. doi: 10.1097/00005792-197707000-00001. No abstract available. PMID 327194
- [Derived] Miao M, Li Y, Huang B, Chen J, Jin Y, Shao M, Zhang X, Sun X, He J, Li Z. Treatment of Active Idiopathic Inflammatory Myopathies by Low-Dose Interleukin-2: A Prospective Cohort Pilot Study. Rheumatol Ther. 2021 Jun;8(2):835-847. doi: 10.1007/s40744-021-00301-3. Epub 2021 Apr 14. PMID 33852146